CLINICAL TRIAL: NCT03529968
Title: Siewert Type I and II Esophageal Adenocarcinoma (EAC): CT, PET-CT, EUS Sensitivity / Specificity for the Assessment of Lymph Node Metastases (LNM) in Groups of Thoracic and Abdominal Lymph Nodal Stations
Brief Title: Siewert Type I-II: CT, PET-CT, EUS Sensitivity/Specificity for the Assessment of Lymph Node Metastases
Acronym: ADECC2-2017
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor, University of Bologna
Other Study IDs: ADECC2-2017
Record Dates: First submitted 2018-04-24; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Siewert Type I-II Adenocarcinoma of the Esophagus
Keywords: esophageal adenocarcinoma; staging; CT; PET-CT; EUS
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Esophagectomy; Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Lymph nodes from surgical samples in patients submitted to surgical procedures for Siwert type I-II esophageal adenocarcinoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Italian Siewert I-II adenocarcinoma: Patients with Siewert type I adenocarcinoma underwent subtotal esophagectomy and proximal gastrectomy with intrathoracic esophagogastric anastomosis. Patients with Siewert type II adenocarcinoma underwent total gastrectomy and esophageal resection at the level of the azygos vein and Roux-en-Y esophagojejunostomy. A right anterolateral thoracotomy and an upper midline laparotomy were performed as previously described. Lymphadenectomy included chest stations classified according to the AJCC TNM 7th edition (L/R = left/right; 3, 4R, 7, 2R, 8 and 9 and abdominal stations classified according to the Japanese Classification of Gastric Carcinoma (stations 1-12)
  Interventions: Procedure: esophagectomy
- Finnish Siewert I-II adenocarcinoma: All Siewert type I/II patients underwent minimally invasive esophagectomy and reconstruction with gastric tube. Laparoscopy and right-sided thoracoscopy in decubitus position were used as previously described. Thoracic lymphadenectomy consisted of stations 7-9 (AJCC TNM 7th edition) and abdominal stations 1-3 and 7-11 according to the Japanese Classification of Gastric carcinoma.
  Interventions: Procedure: esophagectomy

INTERVENTIONS:
Procedure: esophagectomy — Subtotal esophagectomy and proximal gastrectomy with intrathoracic esophagogastric anastomosis. Total gastrectomy and esophageal resection at the level of the azygos vein and Roux-en-Y esophagojejunostomy
  Other Names: gastrectomy

SUMMARY:
In Siewert type I/II EAC, sensitivity/specificity of CT, PET-CT, EUS for assessment of N descriptor in defined groups of lymph nodes were investigated.

DETAILED DESCRIPTION:
Esophageal adenocarcinoma (EAC) is a disease with poor overall prognosis and rising incidence in western countries. In patients without organ metastases, therapy is currently based on surgery with or without neoadjuvant therapy; indication for primary surgery is reserved to clinical TNM stages 0-IIa, whereas a multimodality approach is more suitable for clinical TNM stages IIb-III. The operation comprises the resection of distal esophagus and proximal or total gastrectomy. Two field lymphadenectomy is generally recommended, but the extent of lymphadenectomy is among the controversial issues, as extensive removal of nodes may cause significant morbidity and its effect on survival in addition to neoadjuvant therapy is not clear. Current guidelines are based on the 7th edition of AJCC & UICC TNM classification, which stages lymph node status (N) according to the number of metastatic nodes, but do not consider the specific anatomic stations of regional nodes. EAC subtypes are known to demonstrate different metastatic nodal patterns of spread. They may be classified with the Siewert's classification according to the position of the tumor with respect to the esophago-gastric junction (EGJ), or according to histologic parameters like the presence/absence of intestinal metaplasia in the esophagus and stomach. Siewert Type I EAC, which fairly corresponds to the Barret's like type according to the presence absence of intestinal metaplasia, spreads more likely to the thoracic nodal stations, while Siewert Type II and the pyloric like type, do spread more frequently to the perigastric and celiac stations. Therefore, an increasing interest is emerging for preoperative mapping of lymph nodes metastases in order to tailor surgery according to metastatic patterns.

The majority of studies aiming to assess the accuracy of N staging with clinical methods generally refer to the global evaluation of regional nodes according to the 7th edition of staging descriptors. Studies reporting specific data on the clinical staging assessment of specific thoracic and abdominal lymph nodal stations are few, diagnostic tests and results are not uniform, interpretation and comparison of data within reports is not immediate.

ELIGIBILITY:
Inclusion Criteria:

* Siewert type I-II adenocarcinoma > 18 year submitted to primary surgery

Exclusion Criteria:

* Siewert type I-II adenocarcinoma submitted to neoadjuvant therapy.
* Siewert type III adenocarcinoma Squamous Carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 101 patients affected by Siewert type I (n=60) and type II (n=41) EAC, submitted to up front surgery (no neoadjuvant therapy) in the Thoracic Surgery divisions of the University of Bologna (Maria Cecilia Hospital n=54) and of the Helsinki University Hospital (n=47).
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Principal aim - sensitivity, specificity, accuracy | 1 years
  The aim of this study was to evaluate sensitivity, specificity, accuracy of positron emission tomography integrated with CT (PET-CT), endoscopic ultrasound (EUS) and computed tomography (CT) for staging N descriptor in total (regional N) and in anatomical groups of thoracic and abdominal N stations.
  For each lymph nodal station thoracic and abdominal the outcome measures for CT, PET; EUS were: Sensitivity measured in percentage (number of lymph nodes true positive/number of lymph nodes positive in the test x 100); Specificity measured in percentage (number of lymph nodes true negative/number of lymph nodes negative in the test x 100).

CONTACTS AND LOCATIONS:
Overall Officials: Sandro M Mattioli, MD, Principal Investigator — Department of Medical and Surgical Sciences University of Bologna; Sandro M Mattioli, MD, Study Chair — Department of Medical and Surgical Sciences
Locations (1):
- Department of Medical and Surgical Sciences University of Bologna, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopci E, Kauppi J, Lugaresi M, Mattioli B, Daddi N, Fortunato F, Rasanen J, Mattioli S. Siewert type I and II oesophageal adenocarcinoma: sensitivity/specificity of computed tomography, positron emission tomography and endoscopic ultrasound for assessment of lymph node metastases in groups of thoracic and abdominal lymph node stations. Interact Cardiovasc Thorac Surg. 2019 Apr 1;28(4):518-525. doi: 10.1093/icvts/ivy314. PMID 30496443